CLINICAL TRIAL: NCT05066087
Title: Digital Behavioural Treatment for Improved Functioning and Quality of Life in People With Chronic Pain/ Digital Kognitiv Beteendeterapi för ökad Funktion Och Livskvalitet Hos Personer Med långvarig smärta
Brief Title: Digital Behavioural Treatment for Chronic Pain
Acronym: DAHLIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Linnaeus University (Other); Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Sara Lauren Bartels, Postdoctoral researcher; Principle Investigator, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2021-02437
Record Dates: First submitted 2021-09-06; First posted 2021-10-04 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Focus groups (n=16 patients and n=8 health care professionals); single-arm, iterative sprints with n=10 patients per sprint (total of n=40-60 patients); two-armed RCT with n=180 patients per arm; interviews with stakeholders (minimum of n=6 interviews)
Who Masked: Outcomes Assessor
Masking Description: During the RCT data analysis, the researcher will be blinded (not knowing the participants treatment group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAHLIA treatment (Experimental): 6 weeks of online behavioural treatment; mainly self-guided and weekly contact with their therapist
  Interventions: Behavioral: DAHLIA treatment
- Treatment as usual (Other): receive usual treatment at their rehabilitation centre; detailed information will be collected to define what treatment as usual means in clinical settings.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: DAHLIA treatment — 6 weeks; CBT/ ACT/ process-based treatment; micro-learning format with 4 digital micro-sessions per week; exposure as the core process; guidance to be OPEN, AWARE, ACTIVE; weekly contact with therapist; booster sessions after 2- and 4 months;
  Arms: DAHLIA treatment
Other: Treatment as usual — Usual pain treatment; defined post-hoc based on what patients receive
  Arms: Treatment as usual

SUMMARY:
Overall project aim: to develop, evaluate, and implement a digital behavioural health treatment to improve well-being in individuals with chronic pain.

The treatment will be integrated into the nationally available 1177 web-platform, which will facilitate long-term use in clinical practice across Sweden. Within the project, the investigators will develop the digital treatment and match it to patients' needs using focus groups; pilot the treatment to evaluate its feasibility and acceptability, preliminary efficacy, and individual change processes using the single case experimental design (SCED) method; conduct a two-armed randomized controlled trial enhanced with SCED to assess the clinical effectiveness, cost-effectiveness, and maintenance of change of the treatment compared to treatment as usual; and monitor the implementation process of the treatment through a business model and stakeholder interviews.

DETAILED DESCRIPTION:
Study 1: Identifying and meeting patients' needs Design: Focus groups with individuals with chronic pain and health care professionals. Aim: To identify participant's needs and utilise user input to match the treatment content and design (prototype 1.0) to needs. Sample: People with chronic pain (two focus groups, n=6-8 per group), health care professionals (HCPs) (e.g., psychologists, psychotherapists trained in cognitive behavioural therapy (CBT)) (one focus group, n=6-8) will be recruited from primary care facilities in the region of Kalmar. Data collection: Focus groups will follow a semi-structured guide and be audio- and video-taped. Field notes will furthermore provide insights into relevant cues and observations given by participants. Outcome: Intervention prototype 2.0 Time plan: Autumn/winter 2021.

Study 3: Feasibility, acceptability, preliminary efficacy, and individual change processes Design: Piloting and optimising the treatment in an iterative process with 4-6 smaller cohorts; user input from each optimisation 'sprint' will be integrated and tested in the subsequent cohort/ sprint; single-case experimental design (SCED) method with randomised baseline length, pre- post- and FU-assessment and post-treatment user interviews. Aim: To evaluate the feasibility and acceptability, the preliminary efficacy, and individual change processes of the digital behavioural health treatment within the 1177 web-platform. Sample: People with chronic pain (n=10 per sprint; total of n=60) will be recruited from primary care facilities in the region of Kalmar; the feasibility and acceptability will also be evaluated in treating HCPs (note: one HCP might treat multiple patients at the same time, and also take place in several sprints), who are therefore also considered participants. Data collection: feasibility/ acceptability: semi-structured debriefing interviews of subjective experience combined with objective measures such as drop-out rate, adherence, system-generated technical use e.g. number of log-in time points, number of modules completed; preliminary efficacy: Pre-, post- 3- and 6-month FU-assessment of self-reports on patients' well-being, data of n=60 patients accumulated across all sprints as the treatment remains functionally constant across all optimisation studies; individual change processes: Lunch and evening reports of well-being at least four times per week over the course of the 6-week treatment using a digital diary, also comparing to the baseline and post-treatment diary assessments. Time plan: 2022.

Study 4: RCT enhanced with SCED evaluating the (cost-) effectiveness and maintenance of change Design: Two-armed RCT enhanced with randomized baseline length SCED method comparing the digital behavioural health treatment to primary care treatment as usual (TAU). Aims: To evaluate the clinical effectiveness of the treatment on behavioural health outcomes, and the cost-effectiveness of the treatment in comparison to TAU. Sample: Patients (n=360, n=180 per group) will be recruited from pain clinics and primary care facilities in the region of Kalmar and potentially other regions (e.g., Östergötland, Jönköping, Stockholm, Uppsala, Örebro). Data collection: Self-report questionnaires will be completed over pre-, post- FU-assessments. Furthermore, the digital diary information on daily well-being will be collected at all assessment time points and over the course of the intervention, in both treatment arms. To determine the cost-effectiveness, information from registers on sick leave, medication, and health care consumption will be used . Time plan: 2023-2024.

Study 2 (pre-Implementation) and study 5 (post-implementation): business model, determinants, and lessons-learned Design: Qualitative study using interviews with stakeholders; deductive analysis of qualitative data mapped on the consolidated framework for implementation research. Aim: Identify barriers and facilitators for the prospective implementation of the treatment and prepare the implementation process using a business model canvas (at baseline, study 2); review the actual use and implementation process at follow-up to present lessons learned (at follow-up, study 5). Sample: Various stakeholders identified via snowball-sampling (e.g., development team and facilitators of 1177 web platform at region Kalmar, health care professionals, health care managers, municipality representatives). Interviews will be conducted until data satisfaction is achieved. Data collection: An initial version of a business model canvas will be discussed with the development team and health care managers. Furthermore, potential barriers and facilitators of prospective use will be identified at baseline via a semi-structured interview with the stakeholders. The practical use and implementation status after the treatment is released to the market (here also referred to as follow-up (FU)) will be described using semi-structured interviews to understand the process retrospectively and present lessons learned. Time plan: baseline autumn 2021, FU in autumn 2024 (after RCT, treatment release to other regions).

ELIGIBILITY:
Inclusion criteria

Participant must fulfil the following:

1. be 18 to 65 years of age
2. reporting a pain duration of ≥ 3 months
3. being able to communicate in Swedish
4. having access to a computer, smartphone, and the internet in their home environment.

Exclusion criteria:

Participant may not

1. be injury or illness that require immediate assessment or different treatment, or is expected to progress significantly during the next 6 months
2. taking unstable medication (i.e., changes in medication during the past 3 months or expected within the next 3 months)
3. having received previous CBT treatment (including ACT) during the past 6 months
4. havning severe psychiatric co-morbidity (e.g., high risk of suicide)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change over time in Catastrophizing | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Subscale of coping strategies questionnaire (CSQ), 6-items rated on a 7-point scale, with higher scores indicating higher levels of catastrophizing
Change over time in (Dis)ability/ pain screening | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ), 10 items rated on a 10-point scale, higher scores indicating higher levels of functioning
Change over time in Work ability | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Work ability index (WAI), 10 items rated on different scales (0-10 points, 5-point scale, categorical ratings); no total score but individual information that can be translated into an index or analysed individually
Change over time in Functioning | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Brief pain inventory (BPI-SF), 9 items, question 3-9 rated on a 10-point scale, higher scores indicating greater levels of pain interference

SECONDARY OUTCOMES:
Change over time in Well-being/ depression | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Patient Health Questionnaire (PHQ-9), 10 items rated on a 4-point scale, with higher scores indicating greater levels of depressive symptoms
Change over time in Perceived stress | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Perceived stress scale (PSS), 10 items rated on a 5-point scale, with higher scores indicating greater levels of perceived stress
Change over time in Sleep problems | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Insomnia Severity Index (ISI), 4 items rated on a 5-point scale, with higher scores indicating greater levels of sleeping problems

OTHER OUTCOMES:
Change over time in being Open/ Acceptance | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Chronic Pain Acceptance Questionnaire (CPAQ), 6 items rated on a 7-point scale, with higher scores indicating greater levels of pain acceptance
Change over time in being Aware | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  5 items rated on a 5-point scale, on,'acting with awareness' from the Five Facets MindfulnessQuestionnaire (FFMQ), with greater scores indicating higher levels of awareness
Change over time in being Engaged/ committed action | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  i) Valueing questionnaire (10 items); (ii) Committed action questionnaire (8 items); all items rated on a 7-point scale, with higher scores indicating greater levels of engagement/ committed behaviour
Change over time in Psychological flexibility | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Swedish translation of the Multidimensional psychological flexibility inventory (MPFI), 24 items rated on a 6-point scale with higher scores indicating grater levels of psychological flexibility
Change over time in Self-efficacy | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  general self-efficacy scale (S-GSE), 10 items rated on a 4-point scale, with lower scores indicating greater levels of self-efficacy
Change over time in Pain self-efficacy | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Pain self-efficacy questionnaires (PSEQ-2), 2 items rated on a 7-point scale with higher scores indicating greater levels of pain self-efficacy
Change over time in Avoidance | Pre-post treatment (meaning Baseline and week 7), 3- and 6-month FU
  Avoidance subscale of Psychological Inflexibility in Pain Scale (PIPS), 8 items rated on a 7-point scale with higher scores indicating greater levels of pain-related avoidance

CONTACTS AND LOCATIONS:
Overall Officials: Sara Laureen Bartels, PhD, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Psykisk hälsa, Kalmar
  - Rehab Söder, Kalmar
  - Samrehab, Kalmar
  - Capio St Görans Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
As part of prospective publications, anonymised data will be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol will be published in a scientific journal in 2022. Analytic plans, codes, and data sets will be shared with prospective publications in 2023.
Access Criteria: Data, codes, and plans will be shared through publications. Other researchers may furthermore reach out to get access as a collaboration to additional data sets.

REFERENCES:
- [Derived] Bartels SL, Johnsson SI, Boersma K, Flink I, McCracken LM, Petersson S, Christie HL, Feldman I, Simons LE, Onghena P, Vlaeyen JWS, Wicksell RK. Development, evaluation and implementation of a digital behavioural health treatment for chronic pain: study protocol of the multiphase DAHLIA project. BMJ Open. 2022 Apr 15;12(4):e059152. doi: 10.1136/bmjopen-2021-059152. PMID 35428645
- See also: Research group website — https://ki.se/en/cns/rikard-wicksells-research-group